CLINICAL TRIAL: NCT05871476
Title: Interventions to Decrease Carbapenem Resistant Enterobacteriaceae Colonization and Transmission Between Hospitals, Households, Communities and Domesticated Animals
Brief Title: Interventions to Decrease CRE Colonization and Transmission Between Hospitals, Households, Communities and Domesticated Animals
Acronym: I-CRECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi University of Public Health (Other)
Collaborators: Linkoeping University (Other Government); Karolinska Institutet (Other); Universität Tübingen (Other); University of Copenhagen (Other); National Children's Hospital, Vietnam (Other); Centre de coopération internationale en recherche agronomique pour le développement (CIRAD) (Unknown); International Centre for Antimicrobial Resistance Solutions (Unknown)
Responsible Party: Principal Investigator, Pham-Duc Phuc, Deputy Director of Center for Public Health and Ecosystem Research, Hanoi University of Public Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: JPIAMR 2021-195
Record Dates: First submitted 2023-05-04; First posted 2023-05-23 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Antibiotic Resistant Infection; Carbapenem-Resistant Enterobacteriaceae Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention district (Active Comparator): An information, communication, education and hygiene intervention, developed in collaboration with local health authorities, will aim to improve hygiene and decrease antibiotic use.
  Interventions: Behavioral: , Household Education Communication Hygiene Intervention, Livestock Antibiotic Intervention
- cohort care at the hospital (Active Comparator): A laminated note (yellow for "suspicious CRE carrier": green for (CRE-) patients and red for (CRE+) patients) should be put on the front of the patients' bed.
  Interventions: Behavioral: Hospital Cohort Care Intervention at the hospital

INTERVENTIONS:
Behavioral: Hospital Cohort Care Intervention at the hospital — There will be 3 different cohort groups for the patients: 1) Unknown CRE colonisation status with increased barrier precautions (all patients until screening results arrive will belong to this group unless there are available screening results from referral hospital), 2) CREpos, and 3) CREneg. CREpos patients (2) will be treated in one area of the ICUs by specially assigned nurses/personnel.
  Arms: cohort care at the hospital
Behavioral: , Household Education Communication Hygiene Intervention, Livestock Antibiotic Intervention — The intervention will focus on two main measurable outcomes: 1) Decrease feco-oral-animal transmission route to prevent in-HH and community spread of CRE +/- CoRE. 2) Decrease unindicated community use of ABs for humans and animals. This WP focuses on a one health intervention in collaboration with local health authorities, developing and implementing an HH Education Communication Hygiene Intervention (HECHI) to improve HH hygiene and health management and reduce the risk of transmission between humans and animals, a Provider Engagement Intervention (PEI) to improve case management of common infection and decrease unindicated AB, and and a Livestock AB Intervention (LAI) to reduce the use of AB in livestock through improved biosecurity conditions and animal husbandry.
  Arms: Intervention district

SUMMARY:
Carbapenem resistant Enterobacteriaceae (CRE) colonization of patients discharged from hospitals is a source of transmission to the community. In a cluster randomized controlled trial the effect of a bundle of interventions will be assessed on CRE transmission from CRE+ index patient discharged from hospital to HouseHold (HH) members. The districts in two provinces will be randomized to intervention or control. An information, communication, education and hygiene intervention, developed in collaboration with local health authorities, will aim to improve hygiene and decrease antibiotic (AB) use. The effect will be evaluated on CRE transmission between HH members, livestock and environment through consecutive CRE screening using fecal and hospital effluent samples cultured on carbapenem selective media. Knowledge, Attitudes, Practice surveys with smartphones will assess health seeking, AB use and hygiene adherence, hence detecting the effect of interventions. If transmission of CRE +/- Colistin Resistant Enterobacteriaceae (CoRE, common among livestocks) is detected the source will be investigated including livestock and food, targeted information will be given and evaluated. In hospitals the effect of cohort care will be assessed on CRE acquisition, hospital acquired infection, treatment outcome, costeffectiveness and contamination in sewage water. Mechanisms of resistance, relatedness of CRE isolates in different One Health departments, and rate of CRE transmission from humans to animals and vice versa, will be assessed through Whole Genome Sequencing (WGS).

ELIGIBILITY:
Inclusion Criteria:

* All patients under 2 years old at the selected hospital are highly appreciated to join the study.

Exclusion Criteria:

* Patients not from the selected hospital and individuals outside the selected province

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change the prevalence of CRE colonisation | 12 months from the starting of recruitment patients
  The intervention at hospital will lead to the reduction of CRE colonisation, hospital acquire infection, treatment duration and costs.
Cheng th prevalence of CRE transmission in the household | 12 months from the starting of recruitment community participants
  The Household Education Communication Hygiene Intervention expected to reduce the transmission of CRE from index patient to household member.
Change the awareness regarding AMR of local people | 18 months from the starting of recruitment community participants
  The understanding on AMR, particularly of CRE, proper use of antibiotic for both humans and animals, will be improved. This will be measured through the quantitative questionnaires.
Assessment the effectiveness of the hospital wastewater treatment on reducing CRE from hospital to community | 24 months from the starting of the project
  The presence of CRE in hospital wastewater before and after treatment will be compared to evaluate the effectiveness of the treatment system on preventing the spreading of AMR to the community.
Investigate the genetic relatedness of CRE isolates from hospital, household, animals, wastewater | 24 months from the starting of the project
  The CRE isolated from rectal swab of patient admitted to hospital, household members, animals and wastewater will be subjected to Whole Genome Sequencing using Oxford MinION Nanopore/Illumina Miseq sequencing and bioinformatics analysis to investigate the mechanisms of resistance in different One-Health compartments.

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Larsson, MD, Principal Investigator — Karolinska Institutet; Thirumalaisamy Velavan, PhD, Principal Investigator — University of Tübingen, Germany; Håkan Hanberger, Study Director — Linkoeping University; Flavie Goutard, PhD, Principal Investigator — CIRAD, France; Yaovi Mahuton Gildas Hounmanou, PhD, Principal Investigator — University of Copenhagen; Minh-Dien Tran, Principal Investigator — Vietnam National Children's Hospital
Locations (1):
- Thai Binh Pediatric Hospital, Thái Bình, Thai Binh, Vietnam

IPD SHARING:
Plan to Share IPD: No